CLINICAL TRIAL: NCT00610519
Title: Treatment of Acute Pharyngo-Tonsillitis With Essential Oils of Some Aromatic Medical Plants.
Brief Title: Treatment of Acute Pharyngo-Tonsillitis With Essential Oils of Aromatic Plants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Yoseph Rakover, M.D., Head of Department of Otorhinolaryngology, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: emc070167ctil; Rakover1
Record Dates: First submitted 2008-01-08; First posted 2008-02-08 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Viral Pharyngitis; Viral Tonsillitis
Keywords: Viral pharyngo-tonsillitis;; Herbal medicine;; Traditional medicine;; Aromatic essential oils;

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): treatment with spray containing aromatic essential oils of some herbal plants.
  Interventions: Dietary Supplement: mixture of aromatic essential oils.
- 2 (Placebo Comparator): spray containing placebo.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: mixture of aromatic essential oils. — 3% of mixture containing aromatic essential oils of Eucalyptus citriodora, Eucalyptus globulus, Mentha piperita, Origanum syriacum, and Rosmarinus Officinalis, spraying to the throat.
  Arms: 1
Dietary Supplement: placebo — 0:1% of Lemon VIP (Florasynth,Israel), spraying to the throat.
  Arms: 2

SUMMARY:
This randomized, double blind, parallel group study, compared the efficacy of spray containing aromatic essential oils of some herbal plants, against placebo in the treatment of patients with acute viral Pharyngo-tonsillitis.

Study objectives: Primary to demonstrate a throat pain relief within 20 minutes after first administration of treatment with the spray.

Secondary to demonstrate a reduction of a defined symptoms sum score based on symptoms and signs comparing baseline therapy from the beginning to the end of 3 days treatment

DETAILED DESCRIPTION:
This study compared the efficacy of spray containing aromatic essential oils of Eucalyptus citriodora, Eucalyptus globulus, Mentha piperita, Origanum syriacum, and Rosmarinus Officinalis, against placebo in the treatment of patients with acute viral Pharyngo-tonsillitis.

In- vitro and clinical studies suggest therapeutic potential of aromatic herbs and trees oils in the treatment of Pharyngo-Tonsillitis. The pharmacological and clinical activity of Eucalyptus citriodora, Eucalyptus globulus, Mentha piperita, Origanum syriacum, and Rosmarinus Officinalis, include anti-inflammatory, anti-bacterial and anti-viral activities. Some of these herbs and trees oils have direct activity on the respiratory tract, the coughing reflex and the airflow in the nasal tract.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute viral pharyngo-tonsillitis.
* Active disease less than 48 hours
* Patients agree to sign informed consent according to GCP and Israel national regulations.

Exclusion Criteria:

* Acute follicular tonsillitis.
* Peritonsillar abscess.
* Under any antibiotically treatment.
* Asthma disease.
* Under coumadine therapy.
* Hyper sensitivity to Aromatic essential oils.
* Any immuno-suppressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To demonstrate a throat pain relief within the first 20 minutes after first administration of treatment with the spray. | 20 minutes

SECONDARY OUTCOMES:
To demonstrate a reduction of a defined symptoms sum score based on symptoms and signs comparing baseline therapy from the beginning to the end of 3 days treatment. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Rakover, M.D., Principal Investigator — haemek medical center
Locations (1):
- Otorhinolaryngology department, Afula, Israel